CLINICAL TRIAL: NCT04082364
Title: A Phase 2/3 Trial to Evaluate Margetuximab in Combination With INCMGA00012 and Chemotherapy or MGD013 and Chemotherapy in Patients With Metastatic or Locally Advanced, Treatment-naïve, HER2-Positive Gastric or Gastroesophageal Junction Cancer
Brief Title: Combination Margetuximab, Retifanlimab, Tebotelimab, and Chemotherapy Phase 2/3 Trial in HER2+ Gastric/GEJ Cancer
Acronym: MAHOGANY
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: MacroGenics (Industry)
Collaborators: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGAH22-06
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer; HER2-positive Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — margetuximab; Trastuzumab; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Cohort A is a single-arm cohort to evaluate safety and efficacy of margetuximab plus retifanlimab. Cohort B Part 1 is a randomized, 4-arm segment to evaluate margetuximab plus retifanlimab plus chemotherapy, margetuximab plus tebotelimab plus chemotherapy, margetuximab plus chemotherapy, vs trastuzumab plus chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Chemotherapy-free arm (Experimental): margetuximab plus retifanlimab
  Interventions: Biological: margetuximab; Biological: Retifanlimab
- Margetuximab, retifanlimab, and chemotherapy arm (Experimental): margetuximab plus retifanlimab plus investigator choice of chemotherapy options.
  Chemotherapy options: capecitabine and oxaliplatin (XELOX) or modified 5-FU, leucovorin, and oxaliplatin regimen 6 (mFOLFOX-6)
  Interventions: Biological: margetuximab; Biological: Retifanlimab; Other: Chemotherapy
- Margetuximab, tebotelimab and chemotherapy arm (Experimental): margetuximab plus tebotelimab plus investigator choice of chemotherapy options. Chemotherapy options: capecitabine and oxaliplatin (XELOX) or modified 5-FU, leucovorin, and oxaliplatin regimen 6 (mFOLFOX-6)
  Interventions: Biological: margetuximab; Biological: Tebotelimab; Other: Chemotherapy
- Margetuximab and chemotherapy arm (Experimental): margetuximab plus investigator choice of chemotherapy options. Chemotherapy options: capecitabine and oxaliplatin (XELOX) or modified 5-FU, leucovorin, and oxaliplatin regimen 6 (mFOLFOX-6)
  Interventions: Biological: margetuximab; Other: Chemotherapy
- Trastuzumab and chemotherapy arm (Active Comparator): Trastuzumab plus investigator choice of chemotherapy options. Chemotherapy options: capecitabine and oxaliplatin (XELOX) or modified 5-FU, leucovorin, and oxaliplatin regimen 6 (mFOLFOX-6)
  Interventions: Biological: Trastuzumab; Other: Chemotherapy

INTERVENTIONS:
Biological: margetuximab — margetuximab: Fc-modified anti-HER2 monoclonal antibody: 15 mg/kg IV, Day1 of each 3-week cycle
  Other Names: MGAH22; Margenza®
  Arms: Chemotherapy-free arm; Margetuximab and chemotherapy arm; Margetuximab, retifanlimab, and chemotherapy arm; Margetuximab, tebotelimab and chemotherapy arm
Biological: Retifanlimab — Retifanlimab: anti-PD-1 checkpoint inhibitor 375 mg IV, Day 1 of each 3-week cycle.
  Other Names: MGA012; INCMGA00012
  Arms: Chemotherapy-free arm; Margetuximab, retifanlimab, and chemotherapy arm
Biological: Tebotelimab — Tebotelimab: anti PD-1, anti-LAG3 bispecific DART (R) molecule 600 mg IV, Day 1 of each 3-week cycle.
  Other Names: MGD013
  Arms: Margetuximab, tebotelimab and chemotherapy arm
Biological: Trastuzumab — Anti-HER2 monoclonal antibody 8 mg/kg loading dose and then 6 mg/kg administered IV on Day 1 of each 3-week cycle
  Other Names: Herceptin
  Arms: Trastuzumab and chemotherapy arm
Other: Chemotherapy — Investigator choice of 1 of 2 chemotherapy regimens: XELOX or mFOLFOX6
  Chemotherapy
  XELOX chemotherapy Capecitabine: 1000 mg/m2 as oral capsules twice a day Days 1-14 of each cycle, Oxaliplatin: 130 mg/m2 of Day 1 of each 3-week cycle as IV infusion
  mFOLFOX6 chemotherapy: Leucovorin: 400 mg/m2 every 2 weeks as IV infusion, 5-FU bolus: 400 mg/m2 every 2 weeks as IV infusion, 5-FU continuous infusion: 2400 mg/m2 every 2 weeks as a 46 hr infusion, Oxaliplatin: 85 mg/m2 every 2 weeks as IV infusion.
  Arms: Margetuximab and chemotherapy arm; Margetuximab, retifanlimab, and chemotherapy arm; Margetuximab, tebotelimab and chemotherapy arm; Trastuzumab and chemotherapy arm

SUMMARY:
This is a Phase 2/3, randomized, open-label study for the treatment of patients with HER2-positive Gastric cancer (GC) or Gastroesophageal Junction (GEJ) cancer conducted in two parts.

Part A is a single-arm cohort (Cohort A, 40 to 110 participants) will evaluate safety and efficacy of margetuximab plus retifanlimab.

Part B Part 1 has 4 arms (50 patients/arm). Participants will be randomized to margetuximab plus retifanlimab plus chemotherapy, margetuximab plus tebotelimab, plus chemotherapy, margetuximab plus chemotherapy, or trastuzumab plus chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of previously untreated locally advanced unresectable or metastatic HER2+ GC or GEJ adenocarcinoma

  1. Prior systemic perioperative treatment is allowed; however the participants must have had a disease-free interval of at least 6 months from end of chemo/surgery
  2. Participants receiving perioperative anti-HER2 therapy require testing of HER2 status for eligibility
  3. Cohort A: HER2-positive (by IHC 3+) and PD-L1-positive (by IHC with 22C3 CPS ≥ 1%) per central review
  4. Cohort B: HER2-positive (by IHC 3+ or IHC 2+ in combination with FISH+) by local review. PD -L1 status is not required for enrollment.
* Availability of formalin-fixed, paraffin-embedded tumor specimen, unstained slides or contemporaneous biopsy for tumor target testing
* Eastern Cooperative Oncology Group performance status of 0 or 1, verified within 3 days of Day 1
* Life expectancy ≥ 6 months
* At least one radiographically measurable target lesion
* Acceptable laboratory parameters and adequate organ function

Key Exclusion Criteria:

* Other malignancy that is progressing or required treatment within the past 5 years, with certain exceptions

  * Participants with known MSI-H status
* History of allogeneic stem cell or tissue/solid organ transplant
* Central nervous system metastases
* Clinically significant cardiovascular disease, gastrointestinal disorders, pulmonary compromise

  * Prior neoadjuvant or adjuvant treatment with immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2025-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L. Eck, MD, PhD, Study Director — MacroGenics
Locations (73):
- United States (28):
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center - Duarte, Duarte, California
  - Norris Comprehensive Cancer Center (USC), Los Angeles, California
  - Salinas Memorial, Salinas, California
  - UCLA School of Medicine, Santa Monica, California
  - Yale University, New Haven, Connecticut
  - Florida Cancer Specialists South, Fort Myers, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ocala Oncology Center PL DBA Florida Cancer Affiliates - Ocala, Ocala, Florida
  - Florida Cancer Specialists North, St. Petersburg, Florida
  - Kaiser Permanente, Honolulu, Hawaii
  - University of Chicago, Chicago, Illinois
  - Edward H. Kaplan MD & Associates, Skokie, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Cancer & Hematology Centers of Western Michigan - Lemmen-Holton Cancer Pavilion, Grand Rapids, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Heme Onc, Lincoln, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Stephenson Cancer Center at OUHSC, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Oncology Consultants, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- China (16):
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital (Second People's Hospital Of Jilin Province), Changchun
  - Fujian Medical University - Fujian Provincial Cancer Hospital (Fujian Provincial Tumor Hospital), Fuzhou
  - SIR RUN RUN SHAW Hospital, Zhejiang University school of medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Affiliated Tumor Hospital of Harbin Medical University- the 3rd Affiliated Hospital of Harbin, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Anhui Provincial Cancer Hospital, Hefei
  - Jinan Center Hospital, Jinan
  - Nanjing University Medical School; Nanjing Drug Tower, Nanjing
  - Zhongshan Hospital Fudan University, Shanghai
  - Liaoning cancer hospital, Shenyang
  - Hebei cancer hospital (The Fourth Affiliate), Shijiazhuang
  - Wuhan Union Hospital, Wuhan
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhenzhou
- Germany (4):
  - Institute of Clinical Cancer Research Krankenhaus Nordwest (IKF), Frankfurt
  - Haematologisch-Onkologische Praxis Eppendorf, Hamburg
  - Universitätsmedizin Mainz, Mainz
  - Kliniken Maria Hilf GmbH, Mönchengladbach
- Italy (3):
  - Ospedale San Raffaele, Milan
  - Istituto Europeo Di Oncologia, Milan
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
- Poland (2):
  - SPSK nr 1 in Lublin, Lublin
  - Centrum Medyczne MrukMed, Rzeszów
- Singapore (2):
  - National University Hospital (Cancer Institute) -Singapore, Singapore
  - National Cancer Center Singapore, Singapore
- South Korea (11):
  - Hallym University Sacred Heart Hospital, Anyang-si
  - CHA bundang, Gyeonggi-do
  - Inje University Haeundae Paik Hospital, Haeundae
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Korea University Guro, Seoul
  - Korea University, Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University College of Medicine (Severance Hospital), Seoul
  - Catholic University of Korea St. Vincent Hospital, Suwon
- Taiwan (5):
  - Taipei Medical University Hospital, Taipei City, Taipei
  - Kaohsiung Chang Gung MemorialHospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Keelung, Keelung
  - Liuying Chi MeiMedical Hospital, Tainan
  - National Taiwan University, Taipei
- United Kingdom (2):
  - Cambridge University Hospitals NHS Foundation Trust Addenbrooke's Hospital, Cambridge
  - The Christie Hospital NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Catenacci DV, Rosales M, Chung HC, H Yoon H, Shen L, Moehler M, Kang YK. MAHOGANY: margetuximab combination in HER2+ unresectable/metastatic gastric/gastroesophageal junction adenocarcinoma. Future Oncol. 2021 Apr;17(10):1155-1164. doi: 10.2217/fon-2020-1007. Epub 2020 Dec 2. PMID 33263418

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Chemotherapy-free Arm: margetuximab: 15 mg/kg IV, Day1 of each 3-week cycle Retifanlimab: 375 mg IV, Day 1 of each 3-week cycle.
- Part B: Margetuximab, Retifanlimab, and Chemotherapy Arm: margetuximab: 15 mg/kg IV, Day1 of each 3-week cycle Retifanlimab: 375 mg IV, Day 1 of each 3-week cycle. Chemotherapy: Investigator choice of 1 of 2 chemotherapy regimens: XELOX or mFOLFOX6
- Part B: Margetuximab, Tebotelimab and Chemotherapy Arm: margetuximab: 15 mg/kg IV, Day1 of each 3-week cycle Tebotelimab: 600 mg IV, Day 1 of each 3-week cycle. Chemotherapy: Investigator choice of 1 of 2 chemotherapy regimens: XELOX or mFOLFOX6
- Part B: Margetuximab and Chemotherapy Arm: margetuximab: 15 mg/kg IV, Day1 of each 3-week cycle Chemotherapy: Investigator choice of 1 of 2 chemotherapy regimens: XELOX or mFOLFOX6
- Part B: Trastuzumab and Chemotherapy Arm: Trastuzumab: 8 mg/kg loading dose and then 6 mg/kg administered IV on Day 1 of each 3-week cycle Chemotherapy: Investigator choice of 1 of 2 chemotherapy regimens: XELOX or mFOLFOX6
Period: Overall Study
Arm/Group | Part A: Chemotherapy-free Arm | Part B: Margetuximab, Retifanlimab, and Chemotherapy Arm | Part B: Margetuximab, Tebotelimab and Chemotherapy Arm | Part B: Margetuximab and Chemotherapy Arm | Part B: Trastuzumab and Chemotherapy Arm
Started | 48 | 10 | 6 | 10 | 8
Completed | 17 | 7 | 3 | 2 | 2
Not Completed | 31 | 3 | 3 | 8 | 6
Not completed — Death | 23 | 1 | 1 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 1
Not completed — Follow-up terminated by Sponsor | 5 | 0 | 2 | 3 | 2
Not completed — Disease progression | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Chemotherapy-free Arm: margetuximab: 15 mg/kg IV, Day1 of each 3-week cycle Retifanlimab: 375 mg IV, Day 1 of each 3-week cycle.
- Margetuximab, Retifanlimab, and Chemotherapy Arm: margetuximab: 15 mg/kg IV, Day1 of each 3-week cycle Retifanlimab: 375 mg IV, Day 1 of each 3-week cycle. Chemotherapy: Investigator choice of 1 of 2 chemotherapy regimens: XELOX or mFOLFOX6
- Margetuximab, Tebotelimab and Chemotherapy Arm: margetuximab: 15 mg/kg IV, Day1 of each 3-week cycle Tebotelimab: 600 mg IV, Day 1 of each 3-week cycle. Chemotherapy: Investigator choice of 1 of 2 chemotherapy regimens: XELOX or mFOLFOX6
- Margetuximab and Chemotherapy Arm: margetuximab: 15 mg/kg IV, Day1 of each 3-week cycle Chemotherapy: Investigator choice of 1 of 2 chemotherapy regimens: XELOX or mFOLFOX6
- Trastuzumab and Chemotherapy Arm: Trastuzumab: 8 mg/kg loading dose and then 6 mg/kg administered IV on Day 1 of each 3-week cycle Chemotherapy: Investigator choice of 1 of 2 chemotherapy regimens: XELOX or mFOLFOX6
- Total: Total of all reporting groups
Arm/Group | Chemotherapy-free Arm | Margetuximab, Retifanlimab, and Chemotherapy Arm | Margetuximab, Tebotelimab and Chemotherapy Arm | Margetuximab and Chemotherapy Arm | Trastuzumab and Chemotherapy Arm | Total
Number analyzed (Participants) | 48 | 10 | 6 | 10 | 8 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (12.25) | 61.8 (7.64) | 60.0 (13.45) | 60.5 (13.70) | 61.4 (7.25) | 62.1 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 4 | 1 | 1 | 14
  Male | 42 | 8 | 2 | 9 | 7 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 44 | 10 | 6 | 10 | 8 | 78
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 21 | 10 | 6 | 10 | 8 | 55
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 0 | 0 | 2
  White | 23 | 0 | 0 | 0 | 0 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  South Korea | 19 | 0 | 0 | 0 | 0 | 19
  Singapore | 1 | 0 | 0 | 0 | 0 | 1
  United States | 24 | 0 | 0 | 0 | 0 | 24
  China | 0 | 8 | 5 | 9 | 7 | 29
  Taiwan | 0 | 2 | 1 | 1 | 1 | 5
  Poland | 2 | 0 | 0 | 0 | 0 | 2
  Italy | 1 | 0 | 0 | 0 | 0 | 1
  United Kingdom | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events of Margetuximab Plus Retifanlimab in Cohort A, as Assessed by CTCAE v5.0
Description: Evaluation of adverse events and serious adverse events (Cohort A)
Time Frame: Throughout the study, an average of 11 months.
Population: All patients who receive at least one dose of study drug in Cohort A.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy-free Arm
Number analyzed (Participants) | 48
Participants
  Any AE | 47
  treatment-related AE | 38
  severe AE | 25
  severe treatment-related AE | 12
  AE resulting in whole study treatment withdrawal | 8

2. Primary Outcome: Objective Response Rate (ORR) for Non-microsatellite Instability-high (Non-MSI-H) Participants (Cohort A) Using Investigator-assessed Radiology Reviews
Description: Percent of non MSI-H participants with best overall response of complete response (CR) plus partial response (PR) per RECIST 1.1 (Cohorts A ) based on investigator assessment.
  CR is defined as the disappearance of all target and non-target lesions with no new lesions appearing PR is defined as >= to a 30% decrease in the sum of the longest dimensions of target lesions, non-progression of non- target lesions, with no new lesions appearing.
  CR + PR = ORR
Time Frame: Throughout the study, an average of 11 months.
Population: All participants in Cohort A who received at least one dose of study treatment and had baseline radiographic tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants with CR or PR
Arm/Group | Chemotherapy-free Arm
Number analyzed (Participants) | 48
percentage of participants with CR or PR | 52.1 [37.2 to 66.7]

3. Secondary Outcome: Median Progression-free Survival Using Investigator-assessed Radiology Reviews in Cohort A
Description: Time from start of study treatment to the first documented disease progression per RECIST v1.1 or death due to any cause, whichever occurs first. (Cohorts A) based on investigator assessment
Time Frame: Throughout the study, an average of 11 months.
Population: All participants who were assigned to treatment in Cohort A.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy-free Arm
Number analyzed (Participants) | 48
months | 9.8 [4.60 to 14.75]

4. Secondary Outcome: Median Duration of Response in Cohort A Using Investigator-assessed Radiology Reviews
Description: Time from the date of initial response (CR or PR) to the date of first documented progression or death from any cause, whichever occurs first (Cohorts A)
Time Frame: Throughout the study, an average of 11 months.
Population: All participants in Cohort A who achieved a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy-free Arm
Number analyzed (Participants) | 25
months | 16.1 [9.00 to 21.91]

5. Secondary Outcome: Disease Control Rate
Description: Percentage of patients who experienced response of CR, PR or stable disease for at least 3 months from start of study treatment (Cohorts A and B)
Time Frame: Throughout the study, an average of 11 months.
Population: All participants in Cohort A and B who received at least one dose of study treatment and had baseline radiographic tumor assessment.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Chemotherapy-free Arm | Trastuzumab and Chemotherapy Arm | Margetuximab, Retifanlimab, and Chemotherapy Arm | Margetuximab, Tebotelimab and Chemotherapy Arm | Margetuximab and Chemotherapy Arm
Number analyzed (Participants) | 48 | 8 | 9 | 6 | 10
percent of participants | 83.3 [69.8 to 92.5] | 87.5 [47.3 to 99.7] | 100 [66.4 to 100.0] | 100 [54.1 to 100] | 100 [69.2 to 100]

6. Secondary Outcome: ORR for Cohort B
Description: Proportion of participants with best overall response of CR plus PR per RECIST 1.1
Time Frame: Throughout the study, an average of 11 months.
Population: All participants in Cohort B who received at least one dose of study treatment and had baseline radiographic tumor assessment.
Measure: Number (95% Confidence Interval); unit: percent of participants with CR+PR
Arm/Group | Trastuzumab and Chemotherapy Arm | Margetuximab, Retifanlimab, and Chemotherapy Arm | Margetuximab, Tebotelimab and Chemotherapy Arm | Margetuximab and Chemotherapy Arm
Number analyzed (Participants) | 8 | 9 | 6 | 10
percent of participants with CR+PR | 62.5 [24.5 to 91.5] | 88.9 [51.8 to 99.7] | 83.3 [35.9 to 99.6] | 90.0 [55.5 to 99.7]

7. Secondary Outcome: Number of Participants Who Have Antidrug Antibodies (ADA) to Margetuximab
Time Frame: Throughout the study, an average of 11 months.
Population: Participants in Cohort A and B who received margetuximab as a component of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy-free Arm | Margetuximab, Retifanlimab, and Chemotherapy Arm | Margetuximab, Tebotelimab and Chemotherapy Arm | Margetuximab and Chemotherapy Arm
Number analyzed (Participants) | 48 | 9 | 6 | 10
Participants
  negative at baseline, negative post baseline | 40 | 8 | 5 | 10
  Negative at baseline, positive at least once post baseline | 5 | 1 | 0 | 0
  Positive at baseline, as least once positive post baseline | 2 | 0 | 0 | 0
  Not done at baseline, negative post baseline | 1 | 0 | 0 | 0
  Negative at baseline, not done post baseline | 0 | 0 | 1 | 0

8. Secondary Outcome: Number of Participants Who Have ADA to Retifanlimab
Time Frame: Throughout the study, an average of 11 months.
Population: Participants in Cohort A and B who received retifanlimab as a component of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy-free Arm | Margetuximab, Retifanlimab, and Chemotherapy Arm
Number analyzed (Participants) | 48 | 9
Participants
  negative at baseline, negative post baseline | 43 | 9
  negative at baseline, at least 1 positive post baseline | 3 | 0
  Positive at baseline, and negative post baseline | 1 | 0
  not done at baseline, negative post baseline | 1 | 0

9. Secondary Outcome: Number of Participants Who Have ADA to Tebotelimab
Time Frame: Throughout the study, an average of 11 months.
Population: Participants who received tebotelimab as a component of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Margetuximab, Tebotelimab and Chemotherapy Arm
Number analyzed (Participants) | 6
Participants
  Negative at baseline, negative post baseline | 1
  Negative at baseline, positive at least once post baseline | 4
  negative at baseline, not done post baseline | 1

ADVERSE EVENTS:
Time Frame: AEs are collected from the time of randomization throughout the safety follow up period, an average of 11 months.
Description: AEs are based on physical exam, patient reports, and significant abnormal laboratory values.
  Only patients who received study treatments were assessed for adverse events. Progression of cancer causing hospitalization or death is considered an efficacy outcome and not considered an SAE, unless considered drug-related by the investigator. The protocol-specific definition of an SAE excludes progression of cancer.
Arm/Group | Chemotherapy-free Arm | Margetuximab, Retifanlimab, and Chemotherapy Arm | Margetuximab, Tebotelimab and Chemotherapy Arm | Margetuximab and Chemotherapy Arm | Trastuzumab and Chemotherapy Arm
All-Cause Mortality (participants affected / at risk) | 25/48 | 1/9 | 1/6 | 2/10 | 1/8
Serious Adverse Events (participants affected / at risk) | 20/48 | 4/9 | 5/6 | 4/10 | 2/8
Other Adverse Events (participants affected / at risk) | 47/48 | 9/9 | 6/6 | 10/10 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy-free Arm (N=48) | Margetuximab, Retifanlimab, and Chemotherapy Arm (N=9) | Margetuximab, Tebotelimab and Chemotherapy Arm (N=6) | Margetuximab and Chemotherapy Arm (N=10) | Trastuzumab and Chemotherapy Arm (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 — Low neutrophil count with fever
Thyroiditis subacute (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 — Difficulty swallowing
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 — Painful intestinal obstruction
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 — Gas in the intestinal lining
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 0 | 0 — Fever
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 — Weakness
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 — Gallbladder obstruction
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 — Gallbladder inflammation
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 — Severe bacterial infection
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 — Bladder inflammation
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 — Severe infection
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 — Low potassium in the bloodstream
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 — Low bicarbonate in the blood
Malignant ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Immune-mediated renal disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 — Lung inflammation
Combined pulmonary fibrosis and emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 — An accumulation of fluid around the lungs
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 — A flat red rash with raised areas
Influenza A (Infections and infestations) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy-free Arm (N=48) | Margetuximab, Retifanlimab, and Chemotherapy Arm (N=9) | Margetuximab, Tebotelimab and Chemotherapy Arm (N=6) | Margetuximab and Chemotherapy Arm (N=10) | Trastuzumab and Chemotherapy Arm (N=8)
Anaemia (Blood and lymphatic system disorders) | 14 | 3 | 5 | 9 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 3 | 1 — Low white blood cells
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2 | 0 — Low platelet level
Hypothyroidism (Endocrine disorders) | 5 | 2 | 3 | 0 | 0 — Decreased thyroid function
Diarrhoea (Gastrointestinal disorders) | 18 | 4 | 2 | 4 | 2
Nausea (Gastrointestinal disorders) | 16 | 4 | 1 | 3 | 2
Vomiting (Gastrointestinal disorders) | 16 | 1 | 2 | 3 | 1
Constipation (Gastrointestinal disorders) | 8 | 2 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 10 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 7 | 1 | 0 | 0 | 0 — Indigestion
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 0 — Difficulty swallowing
Fatigue (General disorders) | 14 | 2 | 1 | 0 | 1
Pyrexia (General disorders) | 9 | 0 | 1 | 2 | 1 — Fever
Oedema peripheral (General disorders) | 9 | 0 | 0 | 1 | 1 — Swelling in the extremities
Asthenia (General disorders) | 3 | 0 | 1 | 2 | 0 — Weakness
Chills (General disorders) | 3 | 2 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 4 | 1 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 12 | 3 | 2 | 4 | 1
Platelet count decreased (Investigations) | 3 | 7 | 6 | 7 | 7
Neutrophil count decreased (Investigations) | 1 | 7 | 6 | 10 | 5
White blood cell count decreased (Investigations) | 1 | 7 | 4 | 8 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 6 | 3 | 3 | 4
Alanine aminotransferase increased (Investigations) | 2 | 5 | 0 | 5 | 3
Weight decreased (Investigations) | 9 | 1 | 3 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 2 | 1 | 4 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2 | 2 | 3
Ejection fraction decreased (Investigations) | 3 | 0 | 0 | 2 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 1 | 3 | 1
Blood albumin decreased (Investigations) | 2 | 1 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 2 | 2
Blood creatinine increased (Investigations) | 5 | 0 | 0 | 0 | 0
Protein total decreased (Investigations) | 1 | 1 | 0 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 13 | 3 | 2 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 2 | 4 | 6 | 1 — Decreased albumin in the bloodstream
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 1 | 2 | 3 | 1 — Decreased potassium in the bloodstream
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2 | 3 | 2 | 0 — Decreased sodium in the bloodstream
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 2 | 2 — Decreased calcium in the bloodstream
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 0 | 0 | 0 | 0 — Joint pains
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 2 | 1 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 3 | 1 | 4 | 1
Headache (Nervous system disorders) | 6 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 7 | 1 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 5 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 0 | 0 | 0 — Difficulty breathing
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0 | 0 — Nosebleed
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 1 — Runny nose
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 2 | 1 | 0 | 1 — Itching
Rash (Skin and subcutaneous tissue disorders) | 9 | 1 | 0 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 2 — Redness, pain or swelling of the palms and soles of the feet.
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1 | 0 — A flat red rash with raised areas
Hypertension (Vascular disorders) | 6 | 0 | 0 | 0 | 0 — High blood pressure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT04082364/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT04082364/SAP_001.pdf